CLINICAL TRIAL: NCT00756756
Title: The Effect of Granulocyte Colony Stimulating Factor (G-CSF) on Myocardial Function After Acute Anterior Myocardial Infarction, a Prospective Double Blind Randomized Placebo Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Kojuri J M.D., Shiraz University of medical sciences
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86-3454
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Infarction
Keywords: G-CSF; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): post MI post PCI and G-CSF infusion
  Interventions: Drug: G-CSF
- 2 (Placebo Comparator): post MI and post PCI only placebo infused
  Interventions: Drug: placebo infusion of normal saline

INTERVENTIONS:
Drug: G-CSF — after 2 week post MI an d PCI G-CSF was infused for 5 days at dose of 10 microgram/Kg
  Arms: 1
Drug: placebo infusion of normal saline — 2 week post MI and PCI normal saline was infused
  Arms: 2

SUMMARY:
The investigators applied G-CSF to patients 2 weeks after acute anterior MI and successful PCI to evaluate the efficacy and safety of G-CSF in improving myocardial function as cytokine which improve inflammation and mobilize stem cells from bone marrow for regeneration of myocardium.

DETAILED DESCRIPTION:
Ten patients in the treatment group and 10 patients in the control group were enrolled in this prospective, randomized, double blinded study. Two weeks after myocardial infarction that was accompanied by successful recanalization and stent implantation, the patients of the treatment group received 10 μg/kg body weight per day (divided BID) G-CSF subcutaneously for treatment duration of maximum 5.0 days. In both groups, ejection fraction was evaluated with echocardiography and cardiac scan (Gated SPECT method) 10 days after myocardial infarction and after 6 months. Tei index was measured by echocardiography.

Results: No severe side effects of G-CSF treatment were observed. Ejection fraction determined by cardiac scan increased in the treatment group from 0.428 to 0.462 and from 0.470 to 0.496 in the control group but there was no significant improvement of left ventricular ejection fraction when the G-CSF treated group was compared to the controls (p=0.821 for cardiac scan and p=0.705 for echocardiography). Changes in Tei index was not significant in the treatment group (p=0.815) however it reached significant level in the control group (p=0.005), respectively.

ELIGIBILITY:
Inclusion Criteria:

* First anterior myocardial infarction.
* Low systolic ventricular function.

Exclusion Criteria:

* Bleeding tendency
* Contraindication to G-CSF
* Cardiogenic shock
* Hemodynamic instability
* Hepatic or renal disease
* Multivessel disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 6 months
Diastolic function(Tei index) | 6 months

SECONDARY OUTCOMES:
Drug complication | acute and 6 months
Mortality | 6 months
New revascularization and MACE | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences/Cardiology Ward/Namazi and Shahid Faghihi Hospital, Shiraz, Fars, Iran